CLINICAL TRIAL: NCT03498092
Title: Comparative Study of Bupivacaine Versus Bupivacaine-Dexmedetomidine in Ultrasound Guided Serratus Plane Block for Patients Undergoing Modified Radical Mastectomy
Brief Title: Dexmedetomidine in Serratus Plane Block for Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alaa Mazy (Other)
Responsible Party: Sponsor-Investigator, Alaa Mazy, associate professor of anesthesia and surgical intensive care, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MD/16.06.08
Record Dates: First submitted 2018-04-02; First posted 2018-04-13 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bupivacaine-Dexmedetomidine group (Experimental): After general anesthesia, patients will receive a cocktail of isobaric bupivacaine 2.5 mg/ml plus 5 micrograms (mcg)/ml adrenaline and 1mcg/kg dexmedetomidine in a volume of 0.5 ml/kg injected superficial to serratus muscle between and below latissimus dorsi muscle.
  Interventions: Drug: Bupivacaine-Dexmedetomidine
- Bupivacaine group (Active Comparator): After general anesthesia, patients will receive a cocktail of isobaric bupivacaine 2.5 mg/ml plus 5 micrograms (mcg)/ml adrenaline in a volume of 0.5 ml/kg injected superficial to serratus muscle between and below latissimus dorsi muscle.
  Interventions: Drug: Bupivacaine
- Saline group (Placebo Comparator): This group will serve as a control and blinding group and will receive saline infiltration in the same manner.
  Interventions: Drug: General anesthesia

INTERVENTIONS:
Drug: Bupivacaine-Dexmedetomidine — isobaric bupivacaine 2.5 mg/ml plus 5 micro gram/ml adrenaline and 1 micro gram/kg dexmedetomidine in a volume of 0.5 ml/kg
  Arms: Bupivacaine-Dexmedetomidine group
Drug: Bupivacaine — isobaric bupivacaine 2.5 mg/ml plus 5 micro gram/ml adrenaline in a volume of 0.5 ml/kg
  Arms: Bupivacaine group
Drug: General anesthesia — Normal saline in a volume of 0.5 ml/kg
  Arms: Saline group

SUMMARY:
The serratus plane block (SPB) described by Blanco et al, 2013 is a progression from the work with the Pecs I and II blocks. The serratus muscle is a superficial and easily identified muscle and considered a true landmark to perform thoracic wall blocks because lateral cutaneous branches of the intercostal nerves pierce it in the mid-axillary line. A local anesthetic (LA) is injected under ultrasound (US) guidance either superficial or deep to serratus anterior muscle providing predictable and relatively long-lasting regional anesthesia, which would be suitable for surgical procedures performed on the chest wall.

The linear US probe of frequency (6-13 MHz) is placed over the mid-clavicular region in a sagittal plane.The ribs are counted inferiorly and laterally until the fifth rib in the midaxillary line is identified.The latissimus dorsi, teres major, and serratus muscles are identified.

DETAILED DESCRIPTION:
Possible regional techniques for breast surgery include selective intercostal nerve blockade, thoracic paravertebral blockade, thoracic epidural, intrapleural, local wound infiltration. Each of these techniques has advantages and disadvantages. In general, local or wound infiltration is safe but limited in terms of duration of action, depending on the local anesthetic (LA) used. More invasive techniques such as selective intercostal nerve blocks and thoracic paravertebral blockade may be complicated by pneumothorax or transient Horner's syndrome These techniques are also may be associated with higher risk of local anesthetic toxicity. Besides the neurological side-effects associated with thoracic epidural and paravertebral blocks such as post-sympathectomy hypotension and bradycardia, total spinal block, paraplegia, epidural hematoma, unpredictable spread, intravascular injection also requires special skill precluding their routine use in the setting of day-case surgery. With the use of ultrasound (US) devices in anesthetic practice, newer regional techniques based on detailed knowledge of innervations of the breast are developed as the pectoral nerve (Pecs) block I and II.The breast innervations briefly include lateral and medial pectoral nerves that arise from the brachial plexus innervating the pectoral muscles.The anterior divisions of the thoracic intercostal nerves from T2 to T6. They give off lateral and anterior branches. The Lateral branches pierce the external intercostalis and the serratus anterior muscles at the mid-axillary line to give off anterior and posterior terminal cutaneous branches. The lateral cutaneous branch of the second intercostal nerve does not divide and it is called the intercostobrachial nerve.The Anterior branches pierce the internal intercostalis muscle, the intercostal membranes, and pectoralis major to supply the breast in its medial aspect.The long thoracic nerve passes on the serratus anterior muscle supplying it. The thoracodorsal nerve innervates the latissimus dorsi muscle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of American Society of Anesthesiologists (ASA) grade I - III.
2. Scheduled for unilateral modified radical mastectomy.

Exclusion Criteria:

1. Patient with the skin infection in the axilla.
2. Allergy to local anesthetics of the amide type.
3. Patient refusal.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female patients scheduled for unilateral modified radical mastectomy.
Enrollment: 150 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

PRIMARY OUTCOMES:
The time of the first analgesia request | 24 hours postoperative
  minutes

SECONDARY OUTCOMES:
The total analgesic requirements (Ketorolac) | 24 hours postoperative
  milligram
Pain assessed by Visual Analogue Scale | Postoperative: immediately after surgery, 2, 4, 6,10, 16, 24 hours postoperative
  Visual Analogue Scale: between 0 and 10 (0 representing no pain and 10 is the worst imaginable pain)
Amount of fentanyl consumption | Intraoperative.
  microgram
Mean arterial blood pressure | intraoperative every 30 minutes, and postoperative at 2, 4, 6, 10, 16, 24 hours
  millimeter mercury
Heat rate | intraoperative every 30 minutes, and postoperative at 2, 4, 6, 10, 16, 24 hours
  Beat per minute
Sedation assessed by the observer's assessment of alertness & sedation score | postoperative:10, 20, 30 minutes after extubation
  sedation score (1-5):
  5 = patient respond to name spoken in normal voice.
  4 = patient asleep but arousable to normal tone voice.
  3 = patient asleep but arousable to loud voice.
  2 = patient asleep but arousable by mild prodding or shaking.
  1 = comatose.
The Incidence of postoperative nausea and vomiting | postoperative for 24 hours
  percent
Patient satisfaction assessed by a visual analogue score | postoperative 24 hours after surgery
  A score (0-10): 0 is the least satisfaction,10 the maximum satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Center Mansoura University., Al Mansurah, DKH, Egypt